CLINICAL TRIAL: NCT06665100
Title: Efficacy and Safety of PUL-042 Inhalation Solution in Reducing Lower Respiratory Tract Complications in Patients With Hematologic Malignancies and Recipients of Hematopoietic Stem Cell Transplantation (HSCT) With Documented Viral Infections With PIV, hMPV or RSV
Brief Title: PUL-042 Treatment in Patients With Parainfluenza Virus (PIV), Human Metapneumovirus (hMPV) or Respiratory Syncytial Virus (RSV)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Pulmotect, Inc. (Industry)
Collaborators: Cancer Prevention Research Institute of Texas (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PUL-042-207; CP120014 (Other Grant/Funding Number: Cancer Prevention Research Institute of Texas (CPRIT))
Record Dates: First submitted 2024-10-03; First posted 2024-10-30 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-07

CONDITIONS: Hematologic Malignancies; Hematopoietic Stem Cell Transplant (HSCT)
MeSH Terms: conditions — Hematologic Neoplasms | interventions — Pam2CSK4 acetate and ODN M362 combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- PUL-042 (Experimental): PUL-042 Inhalation Solution
  Interventions: Drug: PUL-042
- Sterile Saline for Inhalation (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PUL-042 — Pam2 : ODN (PUL-042) PUL-042 Inhalation Solution
  Arms: PUL-042
Drug: Placebo — Sterile Saline for Inhalation
  Arms: Sterile Saline for Inhalation

SUMMARY:
The purpose of this research study is to try to see whether an experimental drug, PUL 042 Inhalation Solution (PUL 042), is effective in reducing the severity of lung infections in patients with hematologic malignancies and recipients of hematopoietic stem cell transplantation with documented viral infections due to PIV, hMPV, or RSV. PUL-042 or a placebo will be administered 3 times over a 6-day period. The total duration of the study will be approximately 30 days.

DETAILED DESCRIPTION:
A total of up to 100 participants will be enrolled in this research study, at up to 15 centers. Participants in the study will receive either PUL-042 or a placebo (an inactive agent that appears identical to PUL-042). Patients will be randomized 1:1 for PUL-042 or placebo.

The first 50 patients will either be low dose PUL-042 or placebo. After review of the safety data from the initial patients, the PUL-042 dose may be increased. Subjects will be evaluated by chest x-ray and clinical status for respiratory complications.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be eligible for entry into the study if a nasopharyngeal swab is positive for PIV, RSV, or hMPV (as a single pathogen or a mixed infection with rhinovirus) by molecular assay by a local laboratory AND subjects must fulfill the following inclusion criteria to be eligible for participation in the study:

  1. Subjects with hematologic malignancies (i.e., leukemia, lymphoma, or multiple myeloma) or recipients of an allogeneic or autologous hematopoietic stem cell transplantation for one of the following diagnoses: leukemia, lymphoma, Hodgkin's lymphoma, non-Hodgkin's lymphoma, multiple myeloma, and myelodysplastic and myeloproliferative disorder.
  2. Subjects who have undergone active cytotoxic chemotherapy within 6 months or subjects who are on an immunosuppressive therapy (e.g., alemtuzumab, ibrutinib, mycophenolate mofetil, corticosteroids ≥1mg/kg prednisone equivalent).
  3. Subjects who are recipients of an allogeneic hematopoietic stem cell transplant (HSCT) must be deemed high risk with an Immunodeficiency Scoring Index (ISI) , of greater or equal to 4.
  4. Subjects who are recipients of an autologous HSCT must be within 3 months of the transplant procedure.
  5. Subjects must be symptomatic with upper or lower respiratory tract symptoms such as rhinorrhea, sore throat or cough and must be dosed within 6 days from the onset of symptoms.
  6. Chest X-ray with a Radiologic Severity Index (RSI) score of 6 or lower.
  7. Subjects must have pulse oximetry of hemoglobin saturation ≥ 93% on room air.
  8. Spirometry (forced expiratory volume in one second [FEV1] and forced vital capacity [FVC]) ≥70% of predicted value.
  9. Adult (≥ 18 years of age).
  10. If female, must be either post-menopausal (one year or greater without menses), surgically sterile, or, for female subjects of child-bearing potential who are capable of conception must be: practicing two effective methods of birth control (acceptable methods include intrauterine device, spermicide, barrier, male partner surgical sterilization, and hormonal contraception) during the study and through 30 days after completion of the study. Abstinence is not classified as an effective method of birth control.
  11. If female, must not be pregnant, plan to become pregnant, or nurse a child during the study and through 30 days after completion of the study. A pregnancy test must be negative at the Screening Visit, prior to dosing on Day 1.
  12. If male, must be surgically sterile or willing to practice two effective methods of birth control (acceptable methods include barrier, spermicide, or female partner surgical sterilization) during the study and through 30 days after completion of the study. Abstinence is not classified as an effective method of birth control.
  13. Ability to understand and give informed consent.

Exclusion Criteria:

* Subjects will be excluded if they fulfill any of the following exclusion criteria:

  1. Patients with a pulse oximetry of hemoglobin saturation less than 93% on room air.
  2. Known history of chronic pulmonary disease (e.g., asthma [including atopic asthma, exercise-induced asthma, or asthma triggered by respiratory infection], chronic pulmonary disease, pulmonary fibrosis, COPD), pulmonary hypertension, or heart failure.
  3. Subjects treated for fungal, viral, or bacterial pneumonia in the previous 30 days.
  4. Exposure to any investigational agent (defined as any non-FDA-approved agent) within 30 days, or 5 half-lives of the investigational agent, whichever is longer, prior to the Screening Visit.
  5. Allogeneic HSCT recipients with an ISI of 3 or less.
  6. Autologous HSCT recipients more than 3 months after the transplant procedure.
  7. Patients with a relapsed and/or refractory underlying hematologic malignancy with a life expectancy of less than 2 months.
  8. HSCT recipients in the pre-engraftment period.
  9. Chest X-ray with an RSI of >6.
  10. Patients documented to be positive for other respiratory viruses (limited to influenza, SARS-CoV-2, adenovirus, or coronavirus) within 7 days prior to the Screening Visit, as determined by local testing (additional screening testing is not required).
  11. Clinically significant bacteremia or fungemia within 7 days prior to the Screening Visit that has not been adequately treated, as determined by the Principal Investigator.
  12. Any condition which, in the opinion of the Principal Investigator, would prevent full participation in this trial or would interfere with the evaluation of the trial endpoints.
  13. Previous exposure to PUL-042 Inhalation Solution.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-27 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Efficacy of PUL-042 Inhalation Solution on Lower Respiratory Tract Complications (LRTC) | 28 days
  Determine efficacy of PUL-042 Inhalation Solution on lower respiratory tract complications (LRTC) using the peak post-treatment radiologic severity index (RSI) score in subjects with hematologic malignancies (HM [lymphoma, multiple myeloma and leukemia]) and hematopoietic stem cell transplant (HSCT) recipients with documented parainfluenza virus (PIV), human metapneumovirus (hMPV), or respiratory syncytial virus (RSV) infection. The RSI is a quantitative score based on the presence of pulmonary infiltrates in three zones in both lungs, a total of six zones. Normal in all zones would be a score of zero with a maximum score of 72, which represents total consolidation in all six zones.

SECONDARY OUTCOMES:
Change from Pre-Treatment through 28 days | 28 days
  To determine the difference in the change from pre-treatment to peak post-treatment RSI score through 28 days. The RSI is a quantitative score based on the presence of pulmonary infiltrates in three zones in both lungs, a total of six zones. Normal in all zones would be a score of zero with a maximum score of 72, which represents total consolidation in all six zones.
Proportion of Subjects Positive for Each Virus at Each Sampling Timepoint | 28 days
  To determine the effect of PUL-042 through 28 days for the proportion of subjects positive for each virus at each sampling timepoint.
Change in Viral RNA Shedding Relative to Baseline (copies/mL) | 28 days
  To determine the effect of PUL-042 through 28 days for the change in viral RNA shedding relative to baseline (copies/mL).
Post-Treatment Viral RNA Titers (copies/mL) | 28 days
  To determine the effect of PUL-042 through 28 days for post-treatment viral RNA titers (copies/mL).
Mortality (Incidence) | 28 days
  To determine the effect of PUL-042 through 28 days for mortality (incidence).
Oxygenation Requirements (Days) | 28 days
  The effect of PUL-042 through 28 days on the number of days on supplemental oxygen for each subject.
Duration of ICU Care (Days) | 28 days
  To determine the effect of PUL-042 through 28 days for the duration of ICU care (days).
Incidence of ICU Admission | 28 days
  To determine the effect of PUL-042 through 28 days for the incidence of ICU admission.
Duration of hospitalization (Days) | 28 days
  To determine the effect of PUL-042 through 28 days for the duration of hospitalization (days).
Incidence of Hospitalization | 28 days
  To determine the effect of PUL-042 through 28 days for the incidence of hospitalization.
Respiratory Symptom Scores | 28 days
  To determine the effect of PUL-042 through 28 days for respiratory symptom scores (Patient reported symptoms of cough, shortness of breath, respiratory symptoms [cough + shortness of breath], sputum production and chest pain will each be recorded on a scale of 0 to 3 [0=absent,1= mild, 2= moderate 3= severe]).
Incidence of Pneumonia (Clinical Diagnosis) | 28 days
  To determine the effect of PUL-042 through 28 days (clinical diagnosis).
Adverse Events | 28 days
  To evaluate the incidence and severity of treatment emergent adverse events.
Dose/Response | 28 days
  The efficacy of the 50mcg and 70mcg dose levels relative to placebo on peak RSI and change from baseline in RSI will be calculated and statistical analysis of any difference performed. The RSI is a quantitative score based on the presence of pulmonary infiltrates in three zones in both lungs, a total of six zones. Normal in all zones would be a score of zero with a maximum score of 72, which represents total consolidation in all six zones.

CONTACTS AND LOCATIONS:
Overall Officials: Colin Broom, MD, Principal Investigator — Pulmotect, Inc.
Locations (11):
- United States (11):
  - City of Hope National Medical Center, Duarte, California
  - Northside Hospital, Atlanta, Georgia
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - John Theurer Cancer Center, Hackensack, New Jersey
  - Lineberger Cancer, Chapel Hill, North Carolina
  - OU Health Physicians - Infectious Disease Clinic, Oklahoma City, Oklahoma
  - University of Texas MD Anderson MD Anderson Cancer Center, Houston, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No